CLINICAL TRIAL: NCT03277417
Title: Does the Amniotic Fluid Index Affect the Fetal Cardiac Performance?
Brief Title: Does Amniotic Fluid Index Affect the Fetal Cardiac Performance?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0037-17
Record Dates: First submitted 2017-08-30; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Oligohydramnios; Polyhydramnios
MeSH Terms: conditions — Oligohydramnios; Polyhydramnios

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Isolated Oligohydramnios: Fetuses with amniotic fluid index (AFI) equal or less than 5 cm
  Interventions: Other: Echocardiography
- Isolated Polyhydramnios: Fetuses with amniotic fluid index (AFI) more than 25 cm
  Interventions: Other: Echocardiography
- Control Group: Fetuses with normal amount of amniotic fluid
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Imaging of fetal heart and amniotic fluid

SUMMARY:
To evaluate and compare fetal cardiac performance by fetal echocardiography and delivery outcome between fetuses with isolated oligohydramnios, normal amniotic fluid and polyhydramnios.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24-42 weeks
* Singleton pregnancies

Exclusion Criteria:

* Fetal anatomical or chromosomal abnormality
* Known fetal cardiac defect
* Suspected fetal infection
* Suspected IUGR

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All pregnant women attending the Hillel Yaffe Medical Center's OB/GYN clinic
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Fetal cardiac ventricles | One month
  The width of the fetal cardiac ventricles will be measured and compared between all three groups

SECONDARY OUTCOMES:
Gestational age | One month
  Gestational age at delivery will be compared between the three groups
Mode of delivery | One month
  Mode of delivery will be compared between the three groups
Birth weight | One month
  Birth weight will be compared between the three groups

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Gabbay-Benziv, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No